CLINICAL TRIAL: NCT04527341
Title: Study on Visual Assessment System and Stratified Management Program for Postoperative Delirium After Cardiac Surgery
Brief Title: Postoperative Delirium in Cardiac Surgery ICU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SKQN2020
Record Dates: First submitted 2020-08-23; First posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Delirium
Keywords: postoperative delirium; cardiac surgery; Intensive care unit; risk assessment
MeSH Terms: conditions — Delirium; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cardiac surgery patients in ICU

SUMMARY:
Postoperative Delirium (POD) is a common complication in patients after cardiac surgery, which is associated with short-term prognosis and long-term quality of life. Due to the lack of specific treatment, prevention is the most effective strategy to reduce delirium. Risk assessment greatly contributes to guide prevention by stratifying the risk of the POD. However, the high-quality risk assessment tools are still sparse, and the combination of risk assessment and stratified prevention has not been applied to the management of delirium after cardiac surgery. In the previous work, we found the predictive value of preoperative cardiac function on POD, and found a critical value. On the basis of previous research, this project will learn from previous studies on risk factors of POD, and deeply explore potential predictors. Furthermore, we will develop and validate POD risk prediction model, and then develop it into a visual evaluation system. In addition, based on the theory of risk management and risk assessment tools, using the concepts and methods of evidence-based medicine, the risk assessment system and stratified management program of POD will be formed and evaluated by expert discussion meetings. It is expected that the risk assessment system and stratified management program constructed by this project could simply and quickly screen high-risk patients and carry out timely intervention, so as to reduce the incidence of POD, improve patients' prognosis and the quality of life after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18
* Patients after cardiac surgery
* Admitted to ICU after surgery

Exclusion Criteria:

* Preoperative delirium or dementia patients
* Unable to fully participate in delirium testing, including blind, deaf, illiterate or inability to understand Chinese
* Undergoing surgery procedures do not require admission to SICU
* Transfer to ICU from wards after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged above 18 who are admitted to surgical ICUs after cardiac surgery will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | up to 5 days postoperatively
  Investigators defined patients have delirium if they had at least one positive screening during ICU stay.

SECONDARY OUTCOMES:
Severity of postoperative delirium | up to 5 days postoperatively
  Assess by CAM-ICU-7 if CAM-ICU is positive. Categorized as no delirium: 0-2, mild to moderate delirium: 3-5, and severe delirium: 6-7
duration of postoperative delirium | up to 5 days postoperatively
  Defined as time (in days) from the first positive CAM-ICU until the beginning of two consecutive days of negative CAM-ICU.